CLINICAL TRIAL: NCT03676296
Title: Effect of Puerarin Supplementation on Cardiovascular Disease Risk Factors in Men: a Randomized, Double-blind, Placebo-controlled, 2-way Crossover Trial
Brief Title: Effect of Puerarin on Heart Health in Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Professor Gabriel Matthew Leung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NCD001.0
Record Dates: First submitted 2018-09-11; First posted 2018-09-18 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular Disease Risk Factors
Keywords: Puerarin; Lipids; Testosterone
MeSH Terms: interventions — puerarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puerarin (Experimental): Puerarin (90.2 mg daily) in granules
  Interventions: Drug: Puerarin; Drug: Placebo
- Placebo (Placebo Comparator): Placebo in granules
  Interventions: Drug: Puerarin; Drug: Placebo

INTERVENTIONS:
Drug: Puerarin — Puerarin (90.2 mg daily) in granules (as well as excipients) taken orally for 12 weeks
Drug: Placebo — Placebo in granules (with the same excipients as the puerarin supplement but without puerarin) taken orally for 12 weeks

SUMMARY:
This study aims to assess the effect of puerarin supplementation on cardiovascular disease risk factors in men.

DETAILED DESCRIPTION:
Objectives: To assess the effect of puerarin supplementation on cardiovascular disease risk factors in men.

Study design: A randomized, double-blind, placebo-controlled, 2-way crossover trial of 12-week puerarin supplementation.

Study subjects: 234 Hong Kong Chinese men aged 18-50 years without a history of cardiovascular disease.

Intervention: After assessing eligibility, all participants will be randomized to take a puerarin supplement in granules (90.2 mg daily) or a placebo, followed by a 4-week wash-out period, after which participants will be crossed over to the other intervention.

Primary outcomes: Lipid profile (total cholesterol, low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol, triglycerides).

Secondary outcomes: Cardiovascular disease risk factors, such as blood pressure and fasting glucose, as well as some potential mediating pathways, such as testosterone.

Methods: An intention to treat analysis will be used, assuming no changes in baseline value for missing follow up values. Differences in outcomes between supplementation and placebo within participants will be compared using a paired t-test, after checking for the possibility of a carryover effect.

Expected results: The short-term effect of puerarin on cardiovascular disease risk factors in men will be obtained so as to confirm or refute previous trials usually with small sample sizes that suggest puerarin may improve lipid profile and reduce testosterone. The findings will also add evidence about the effects of puerarin on other potentially relevant risk factors, such as blood pressure, fasting glucose and testosterone, as well as some related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Aged 18 to 50 years
* Chinese ethnicity
* Willing to make return visits
* Not currently taking any traditional Chinese medicine (including puerarin) supplementation
* Not currently receiving hormone replacement therapy, such as testosterone replacement therapy, in the past 12 months
* Free of any congenital diseases
* Free of any infectious diseases e.g. seasonal influenza
* With no history of any chronic diseases including coronary heart disease (ischemic heart disease), myocardial infarction (heart attack), stroke, diabetes and cancer
* Have a 10-year risk of ischemic heart disease of less than 10%

Exclusion Criteria:

* Women
* Men, who did not meet the aforementioned inclusion criteria, and/or unable or unwilling to provide consent

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
Change in total cholesterol | Baseline, 12 weeks, 16 weeks and 28 weeks
  Mean difference in total cholesterol (mmol/L)
Change in low density lipoprotein (LDL) cholesterol | Baseline, 12 weeks, 16 weeks and 28 weeks
  Mean difference in LDL cholesterol (mmol/L)
Change in high density lipoprotein (HDL) cholesterol | Baseline, 12 weeks, 16 weeks and 28 weeks
  Mean difference in HDL cholesterol (mmol/L)
Change in triglycerides | Baseline, 12 weeks, 16 weeks and 28 weeks
  Mean difference in triglycerides (mmol/L)

SECONDARY OUTCOMES:
Change in blood pressure | Baseline, 12 weeks, 16 weeks and 28 weeks
  Mean difference in systolic and diastolic blood pressure (mmHg)
Change in fasting glucose | Baseline, 12 weeks, 16 weeks and 28 weeks
  Mean difference in fasting glucose (mmol/L), with log transformation if appropriate
Change in testosterone | Baseline, 12 weeks, 16 weeks and 28 weeks
  Mean difference in testosterone (nmol/L), with log transformation if appropriate

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel M Leung, M.D., Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No